CLINICAL TRIAL: NCT03479255
Title: Smartphone-Enabled Supervised Exercise Therapy for the Treatment of Symptomatic Peripheral Arterial Disease
Brief Title: Smartstep Smartphone PAD
Acronym: SMARTSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Woodruff Health Sciences Center Foundation (Unknown)
Responsible Party: Principal Investigator, Amit J. Shah, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00102543
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Smartphone; Exercise; Functional capacity
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective clinical trial that will randomize patients in 1:1 ratio to smartphone-enabled structured exercise therapy (SE-SET) vs. standard exercise therapy (usual care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smartphone-enabled structured exercise therapy (SE-SET) (Experimental): This arm involves a smartphone app Movn - rehabilitation platform based on MULTIFIT, a case-management system for secondary prevention and patient surveillance after acute MI.
  The key features of the smartphone app include daily reminders to exercise, virtual diary for patients to enter data on exercise sessions, two-way secure messaging with the health coach, and educational videos on heart and vascular health.
  Interventions: Behavioral: Smartphone-enabled structured exercise therapy (SE-SET)
- Standard exercise therapy (Active Comparator): Self-directed, unsupervised exercise as prescribed by the patient's physician.
  Interventions: Behavioral: Standard exercise therapy

INTERVENTIONS:
Behavioral: Smartphone-enabled structured exercise therapy (SE-SET) — The SE-SET program lasts a total of 12 weeks per participant. During this time, the application will automatically track physical activity (steps) and subjects will be prompted to enter other health data such as blood pressure and weight and watch brief educational videos on topics such as smoking cessation, low sodium diet, high fruit/vegetable intake, and medication adherence/education. Patients will be contacted by a member of the study team weekly via phone call to identify barriers to patient compliance (issues related to exercise tracking, medication issues that prevent patients from being active, high BP/weight issues) and help patients navigate those barriers. Movn participants can also send direct messages to the study team to ask about non-urgent matters related to their care.
  Arms: Smartphone-enabled structured exercise therapy (SE-SET)
Behavioral: Standard exercise therapy — The Standard exercise therapy lasts a total of 12 weeks per participant. Participants will be counseled by the physician to perform exercise at home, including 3 times per week of walking 30+ minutes; if applicable, the physician will also counsel on smoking cessation, low sodium diet, high fruit/vegetable intake, and medication adherence/education. These patients will be given a fitness band, which will be set up by the study team using a de-identified study account that will provide additional data on their progress over time.
  Arms: Standard exercise therapy

SUMMARY:
The study aim is to evaluate the effectiveness of a coached, smartphone-enabled exercise program versus physician directed exercise therapy (usual care).

DETAILED DESCRIPTION:
Structured exercise therapy is a first line treatment for symptomatic peripheral artery disease, but compliance is poor. Coaching programs may help but requires significant resources. Smartphone programs may increase the efficiency of such efforts. The study aim is to evaluate the effectiveness of a coached, smartphone-enabled exercise program versus physician directed exercise therapy (usual care) in patients at Grady Memorial Hospital's vascular clinic.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable intermittent claudication
* Able to give informed consent
* Age 18-89 years

And one of the following:

* ABI < 0.9 after 10 minutes of rest OR
* For subjects with an ABI of >1.3 (non-compressible arteries) a Toe-Brachial Index (TBI) of < 0.70 must be obtained for subject qualification. If ABI is > 0.9 to 1.0, a reduction of 20% in ABI must be measured within 1 minute of treadmill testing.

Exclusion Criteria:

Life-threatening process including:

* Sepsis
* Critical limb ischemia (Rutherford class 4-6)
* Unstable angina
* Active malignancy with life expectancy < 6 months
* Severe NYHA Class IV heart failure

Condition other than PAD that limits walking before claudication onset

This includes, but is not limited to:

* Severe angina or dyspnea
* Arthritis
* Muscle weakness/pain

Active behavioral conditions such as uncontrolled schizophrenia or illicit drug addiction that, in the opinion of the study team, will interfere with active participation

Inability to attend study visits

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk test (6MWT) distance completed | Immediately before and after the 12-week period
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

SECONDARY OUTCOMES:
Change in Walking Impairment Questionnaire (WIQ) score | Immediately before and after the 12-week period
  WIQ measures self-reported walking distance, speed, and stair-climbing ability. In the WIQ distance score, the participant is asked to assess the degree of walking difficulty in walking specific distances on a scale from 0 to 4. A score of 0 represents the inability to walk the distance and a score of 4 represents no difficulty. WIQ speed score assesses the degree of difficulty in walking one block at specific speeds, ranging from walking slowly to jogging, on a scale of 0 to 4. In the WIQ stair-climbing score, the participant is asked to report the degree of difficulty climbing specific numbers of flights of stairs, ranging from one to three flights of stairs, on a scale of 0 to 4. This graded score is multiplied by a prespecified weight for each distance, speed, or number of stair flights. The products are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform any of the tasks) to 100 (representing no difficulty).
Change in Physical Health Composite Score of SF-36 | Immediately before and after the 12-week period
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to use special software. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.
Change in claudication onset time during 6MWT | Immediately before and after the 12-week period
  One typical symptom of peripheral arterial occlusive disease' (PAOD) is claudication , which is defined as pain, cramps, numbness or a sense of fatigue in the muscles associated with walking, in one or both lower limbs, affecting either the distal or proximal muscle groups.
Change in ankle-brachial pressure index (ABPI) | Immediately before and after the 12-week period
  The ankle-brachial pressure index (ABPI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). Compared to the arm, lower blood pressure in the leg suggests blocked arteries due to peripheral artery disease (PAD). The ABPI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm.
Change in number of steps/week | Immediately before and after the 12-week period
  Number of steps/week will be obtained from participants' fitness trackers
Critical Limb Ischemia | Over the 12-week study period
  Number of Critical Limb Ischemia events reported by participants
Other Cardiovascular Outcomes | Over the 12-week study period
  Number of Cardiovascular Outcomes other than Critical Limb Ischemia events reported by participants
Exercise-Related Injury | Over the 12-week study period
  Number of Exercise-Related Injury events reported by participants
Mortality | Over the 12-week study period
  Number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Amit Shah, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System (non-CRN), Atlanta, Georgia, United States